CLINICAL TRIAL: NCT04811222
Title: Gallium-DOTATATE PET-MR Imaging to Detect Macrophages in Abdominal Aortic Aneurysms
Brief Title: DOTATATE PETMRI AAA Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-5802
Record Dates: First submitted 2021-03-10; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: Ga-DOTATATE PETMRI scan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ga-DOTATATE PET/MRI scan (Experimental): Patients with abdominal aortic aneurysm will undergo Ga-DOTATATE PET/MRI scan
  Interventions: Diagnostic Test: Ga-DOTATATE PETMRI scan

INTERVENTIONS:
Diagnostic Test: Ga-DOTATATE PETMRI scan — Patients with AAA with minimum 2 years surveillance will have one time Ga-DOTATATE PETMRI scan

SUMMARY:
Abdominal Aortic Aneurysm (AAA) screening and an aging population have increased the prevalence of AAA diagnoses. Small AAAs (<5.5cm) are monitored with ultrasound. Large AAAs may rupture and this is usually fatal. Surgery is considered at a crude size threshold of 5.5cm when the annual rupture risk reaches 5%. AAA size is the only predictor of growth and rupture available but growth is non-linear and some small AAAs rupture. Thus, only 1 in 20 patients treated at 5.5cm will have benefited from rupture prevention in the year following surgery, and others may miss out on life-saving surgery. This study will develop an imaging tool PETMRI with radiotracer Ga- DOTATATE with high clinical utility, to improve prediction of aneurysm growth and risk.

DETAILED DESCRIPTION:
The prevalence of abdominal aortic aneurysm (AAA) in those over 65 years is 4-8% and rising. Currently, AAA size is the only metric to determine risk of growth/rupture; we are unable to image the underlying disease process. Using size alone is problematic. For small AAAs there is no consensus between surgical societies on appropriate surveillance intervals. AAA growth is non-linear and thus some small AAAs may rupture between screening intervals.

Macrophage mediated inflammation leads to weakening of the aortic wall. Our own laboratory work indicates macrophages correlate with AAA severity in mice. In humans, activated macrophages express SomatoSTatin Receptor 2 (SSTR2). For the first time ever, using a radiotracer probe specific for SSTR 2 (gallium-dotatate), we will detect activated macrophages in AAAs using Positron Emission Tomography- Magnetic Resonance Imaging (PET-MRI). Patients attending the University Health Network (UHN) Vascular clinic undergoing ultrasound surveillance of small AAAs of differing sizes will be imaged with Ga-Dotatate PET-MRI. We will correlate aneurysm size and anatomical information with in-vivo imaging of aortic macrophages detected with Ga-Dotatate, to determine the risk of aneurysm growth.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of asymptomatic abdominal aortic aneurysm AAA >3cm in maximum diameter;
2. Minimum 2 years prior ultrasound or CT imaging of their AAA;
3. No prior treatment for AAA;
4. Age >50 years;
5. No contraindications to PET/MRI, such as claustrophobia;

Exclusion Criteria:

1. Pregnant females. All women of child-bearing potential must receive a negative urine pregnancy test prior to administration of 68Ga-DOTATATE;
2. Allergy and/or hypersensitivity to MRI contrast agents (gadolinium) or components of 68Ga-DOTATATE drug product (as listed in IB);
3. Presence of pacemaker or implanted cardioverter defibrillator (ICD);
4. History of alcohol or substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
68-Ga DOTATATE uptake | within 6 months after obtaining consent
  Measuring AAA patient's 68-Ga DOTATATE uptake using PET/MRI as a marker of macrophage accumulation

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Veit-Haibach, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada